CLINICAL TRIAL: NCT04900220
Title: Investigating Differences in Flare Reaction Incidence and Intensity Following Trigger Finger Injections Using Betamethasone and Methylprednisolone
Brief Title: Differences in Flare Reaction Incidence and Intensity Following Trigger Finger Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Shafic Sraj, MD, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2103263450
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Results first posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-05

CONDITIONS: Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Betamethasone; Methylprednisolone

STUDY DESIGN:
Intervention Model Description: This is a double-blinded randomized trial enrolling patients into one of the two treatment groups. The volume of the doses of steroid to be given will be standardized to 1 cc of either methylprednisolone (40 mg) or betamethasone (6 mg). We will instruct patients who meet the inclusion criteria to complete a visual analog scale (VAS) of their pain (1-10) prior to the injection, immediately after the injection, five minutes after the injection, and once a day for a minimum of 7 days after the injection. The incidence, intensity, time to peak and time to resolution of the flare reactions (defined as a 2-point increase from pre-injection pain) will be assessed and compared between the two groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Betamethasone (Active Comparator): betamethasone
  Interventions: Drug: Betamethasone
- Methylprednisolone (Active Comparator): methylprednisolone
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Betamethasone — The volume of the doses of steroid to be given will be standardized to 1 injection of 1 cc of betamethasone (6 mg)
  Arms: Betamethasone
Drug: Methylprednisolone — The volume of the doses of steroid to be given will be standardized to 1 injection of 1 cc of methylprednisolone (40 mg)
  Arms: Methylprednisolone

SUMMARY:
Two common corticosteroids used for trigger finger treatment are betamethasone and methylprednisolone. Both injections are effective in treating trigger finger and the decision of which to use in treatment is currently a matter of the current practice and physician preference. The goal through this randomized trial is to see whether there is a difference between these two corticosteroids in inducing flare reactions and if there are any differences in the peak level of pain and their duration. Findings indicating a statistically significant difference in the incidence and/or intensity of the flare reactions would be clinically significant and would be evidence supporting the switch of current practice to one corticosteroid over the other.

DETAILED DESCRIPTION:
Corticosteroid injections are effective non-surgical approach to treating trigger finger (stenosing tenosynovitis) with success rates reported as high as 92% after just one injection [1]. Among their side effects is a post-injection flare of increased pain that is attributed to crystal-induced synovitis. Reports of these flares in the literature have been rare. Recent evidence their incidence can be as high as 33%. The investigators feel it is a more common clinical issue than traditionally reported and it would be beneficial to control and reduce their incidence if possible.

Two common corticosteroids used for trigger finger treatment are betamethasone and methylprednisolone. Both injections are effective in treating trigger finger and the decision of which to use in treatment is currently a matter of the current practice and physician preference. There is no literature comparing the side effects, specifically flare reactions between these two treatments. The goal through this randomized trial is to see whether there is a difference between these two corticosteroids in inducing flare reactions and if there are any differences in the peak level of pain and their duration.

This is a double-blinded randomized trial enrolling patients into one of the two treatment groups. The volume of the doses will be standardized to 1 cc of either methylprednisolone (40 mg) or betamethasone (6 mg). Patients, who meet the inclusion criteria, will be instructed to complete a visual analog scale (VAS) of their pain (1-10) prior to the injection, during the injection and once a day for the following 7 days after the injection. The investigators estimate that a minimum of 30 patients in each group will be needed to achieve a minimum of 80% power and 0.05 significance. The incidence, intensity, time to peak and time to resolution of the flare reactions (defined as a 2-point increase from pre-injection pain) will be assessed and compared between the two groups. Findings indicating a statistically significant difference in the incidence and/or intensity of the flare reactions would be clinically significant and would be evidence supporting the switch of current practice to one corticosteroid over the other.

ELIGIBILITY:
Inclusion Criteria:

* Single trigger injection
* First time for the digit
* No prior surgery on digit

Exclusion Criteria:

* Current oral steroid use
* Rheumatoid arthritis
* More than one single digit involved
* Previous injection in same digit
* Prior surgery on same digit
* Other injections in the same clinic on the same day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2023-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shatic Sraj, MD, Principal Investigator — West Virginia University
Locations (2):
- United States (2):
  - WVU Medicine University Town Center, Morgantown, West Virginia
  - Ruby Memorial Hospital or Other WVU Healthcare Site, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients seen in the Hand Clinic for single trigger finger issues were approached for the project.
Period: Overall Study
Arm/Group | Betamethasone | Methylprednisolone
Started | 33 | 33
Completed | 32 | 32
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Betamethasone | Methylprednisolone | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (12.7) | 58.5 (12.6) | 60.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 23 | 41
  Male | 14 | 9 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64
Tobacco Use [Count of Participants; unit: Participants]
  Smokers | 4 | 2 | 6
  Non-Smokers | 28 | 30 | 58
Hand Dominance [Count of Participants; unit: Participants]
  Right | 29 | 27 | 56
  Left | 3 | 5 | 8
Side of Trigger [Count of Participants; unit: Participants]
  Right | 20 | 20 | 40
  Left | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Pain
Description: Recorded when subject reports pain. Assessed using the visual analog scale (0-10 scale). Zero indicates no pain, 10 indicates worst pain ever
Time Frame: Up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Methylprednisolone
Number analyzed (Participants) | 32 | 32
Participants | 6 | 11

2. Primary Outcome: Intensity of Pain
Description: Assessed using the visual analog scale (0-10 scale). Zero indicates no pain, 10 indicates worst pain ever
Time Frame: Up to 7 days
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Betamethasone | Methylprednisolone
Number analyzed (Participants) | 32 | 32
score on a scale
  Baseline | 2.8 [0 to 10] | 2.1 [0 to 10]
  Five Minutes | 0.3 [0 to 10] | 0.8 [0 to 10]
  Day 1 | 1.4 [0 to 10] | 2.9 [0 to 10]
  Day 2 | 1.3 [0 to 10] | 2.1 [0 to 10]
  Day 3 | 1.0 [0 to 10] | 1.5 [0 to 10]
  Day 4 | 0.7 [0 to 10] | 1.0 [0 to 10]
  Day 5 | 0.6 [0 to 10] | 0.8 [0 to 10]
  Day 6 | 0.6 [0 to 10] | 0.7 [0 to 10]
  Day 7 | 0.5 [0 to 10] | 0.6 [0 to 10]

3. Primary Outcome: Incidence of Flare Reaction
Description: Number of patients having a severe flare reaction
Time Frame: From baseline up to 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Betamethasone | Methylprednisolone
Number analyzed (Participants) | 32 | 32
Participants
  Severe Flare | 2 | 5
  No Severe Flare | 30 | 27

ADVERSE EVENTS:
Time Frame: Adverse events were reviewed over a 7 day period, from time of injection until flare resolution.
Arm/Group | Betamethasone | Methylprednisolone
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT04900220/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT04900220/ICF_001.pdf